CLINICAL TRIAL: NCT04893590
Title: Adapting MHealth Technology to Improve Patient Activation and Overall Wellness for Persons with Disabilities
Brief Title: Adapting MHealth Technology to Improve Patient Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupation Therapy and Neurology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202103191
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Stroke; Multiple Sclerosis
Keywords: Fatigue; Persons with disabilities; Patient activation; Mobile health
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Multiple Sclerosis; Fatigue; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fatigue self-management SMS intervention (Experimental): The participants will receive a 12-week fatigue self-management SMS text intervention using mobile phones to target patient activation levels in people with disabilities.
  Interventions: Behavioral: Fatigue self-management SMS intervention

INTERVENTIONS:
Behavioral: Fatigue self-management SMS intervention — Participants will set up an initial goal for the SMS intervention related to fatigue management, and prior to beginning the intervention they will be trained to use the SMS system. Participants will receive text messages each day, providing tips and techniques to help self-manage fatigue. Weekly the participants will be asked to provide feedback regarding their fatigue levels and their patient activation will be re-assessed at the halfway point of intervention.

SUMMARY:
Persons with disabilities (PwD) commonly experience fatigue, which often negatively impacts their everyday lives. Management of this symptom can be challenging. Satisfaction with current interventions to manage fatigue is low among PwD and there is a desire for more personalized approaches. The purpose of this study is to develop and test a fatigue self-management intervention using mobile phones that is personalized to each person's needs.

DETAILED DESCRIPTION:
Persons with disabilities (PwD) commonly experience fatigue, which adversely impacts their everyday lives. Information to manage and improve fatigue can be complicated and overwhelming. Little has been done to link mobile health (mHealth) approaches with patient activation and self-management to effectively address fatigue for PwD. The purpose of this study is to develop and pilot-test a fatigue self-management short message service (SMS) text intervention using mobile phones to target patient activation levels in PwD. The proposed study will: (1) develop content for a fatigue self-management intervention using SMS tailored to patient activation levels in persons with multiple sclerosis, spinal cord injury, and stroke. An advisory board made up of one physical medicine and rehabilitation physician and six PwD will provide input on the content and format for the developed content. (2) test the feasibility and acceptability of SMS to improve patient activation for fatigue self-management in PwD. The long-term goal is to improve the health of PwD by increasing their skills, confidence, and knowledge to manage fatigue and other chronic symptoms that affect their daily life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* had disability for at least one year
* score of less than 10 on the Modified Fatigue Impact Scale 5 question (MFIS-5)
* ability to read and speak English at the 6th grade level
* willing to use their own phone and SMS

Exclusion Criteria:

* evidence of acute condition (e.g. relapse)
* sleep apnea
* inability to answer interview questions or provide consent
* terminal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Patient Activation - change in knowledge, skill and confidence for self-management | Baseline and up to 2 weeks post intervention
  The Patient Activation Measure (PAM-13) assesses four levels of activation: (1) the patient is disengaged and overwhelmed, (2) the patient is becoming aware but still struggling, (3) the patient takes action, and (4) the patient maintains behaviors. The psychometric properties of the PAM have been assessed in multiple healthcare settings. Raw PAM scores can be transformed into a continuous (0-100) scale, where higher scores represent higher levels of patient activation. In order to target self-management strategies, participants will proceed through these levels.

SECONDARY OUTCOMES:
The Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue Short Form 8a | Baseline and up to 2 weeks post intervention
  The Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue and the impact of fatigue. The fatigue short forms are not disease specific and assess fatigue over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
The Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Short Form 8a | Baseline and up to 2 weeks post intervention
  The Sleep disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. The sleep disturbance short forms are not disease specific and assess sleep disturbances over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "very poor (1)" to "very good (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States